CLINICAL TRIAL: NCT04272931
Title: DRAGON 1- Training, Accreditation, Implementation and Safety Evaluation of Portal and Hepatic Vein Embolization to Accelerate Future Liver Remnant (FLR) Hypertrophy
Brief Title: DRAGON 1- Training, Accreditation, Implementation and Safety Evaluation of Combined PVE/HVE
Acronym: DRAGON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Maastricht University (Other)
Collaborators: Koningin Wilhelmina Fonds (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL71535.068.19
Record Dates: First submitted 2020-01-07; First posted 2020-02-17 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Colorectal Cancer Liver Metastases
Keywords: Future Liver Remnant; Portal and Hepatic Vein Embolization; Colorectal Liver Metastases

STUDY DESIGN:
Intervention Model Description: Multicenter, international, prospective, multi-center trial to test enrolment capacity of participants and safety of Portal and Hepatic Vein Embolization (PVE/HVE): DRAGON 1 will form the basis of a planned subsequent trial ("DRAGON 2") that will compare PVE with PVE/HVE. In DRAGON 1 every center has to demonstrate the ability to enroll 3 patients in 12 months safely
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Portal and Hepatic Vein Embolization (Experimental): 3 patients per center over one year approximately 90 patients in total. Patients will undergo portal vein and hepatic vein embolization instead of only portal vein embolization.
  Interventions: Procedure: Portal and Hepatic Vein Embolization

INTERVENTIONS:
Procedure: Portal and Hepatic Vein Embolization — Procedure/Surgery: Combined portal vein embolization and hepatic vein embolization (PVE/HVE) • All techniques of PVE allowed (ipsi-lateral, contra-lateral, trans-splenic, all embolization agents except for ethanol alone) • All modifications of HVE allowed (venous occlusion umbrellas; trans-jugular, trans-hepatic, no use of vein glue to avoid lung embolization; staged approach allowed, but first PVE, then HVE and within 48 hours)
  Other Names: Liver venous deprivation (LVD); Double embolization

SUMMARY:
Brief Summary: Some colorectal liver metastases can only be resected after inducing liver regeneration by portal vein embolization (PVE) to increase size function of the future liver remnant (FLR). While PVE is standard, embolization of portal vein and hepatic veins (PVE/HVE) on one side of the liver may faster and more extensive liver size and function growth. PVE/HVE is a novel procedure and requires a safety and feasibility evaluation in a pretrial (DRAGON1) to then be compared in a randomized controlled trial (RCT) to PVE (DRAGON 2).

DETAILED DESCRIPTION:
Detailed Description: Resection of liver metastases from colorectal cancer (CRLM) improves survival compared to chemotherapy alone and may lead to cure in up to 40% of patients. Surgical resectability is limited by location of metastases and by FLR size and function. Commonly, the volume of the future liver remnant (FLR) should be at least 30% of the functional FLR volume. If this volume criterion is not met, the induction of liver regeneration between a two-stage hepatectomy is performed at many centers, with the aim to render patients resectable and reduce the risk of post hepatectomy liver failure. Gold standard to induce regeneration is the embolization of the portal vein branches to the tumor carrying liver (PVE) to induce regeneration of the FLR. Recently, combined embolization of both portal and hepatic veins (PVE/HVE) has been described as an alternative to portal vein embolization because it accelerates and increases growth of the FLR. PVE/HVE combines simultaneous embolization of the portal main branches into the tumor bearing liver and the hepatic vein draining them. The tissue in the part of the liver treated with PVE/HVE stays viable because the hepatic artery continues to supplies the liver deprived of portal and hepatic veins. Preclinical studies in pigs have demonstrated feasibility of this method and human case series show accelerated and increased liver growth. No multi-center evaluation has been performed so far. DRAGON 1 is an international, prospective, multi-center trial to test enrolment capacity of participants and safety of portal and hepatic vein embolization (PVE/HVE). DRAGON 1 will form the basis of the RCT DRAGON 2 to compare PVE with PVE/HV. DRAGON 2 is expected to start in 2021.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primarily unresectable/potentially resectable CRLM after conversion chemotherapy with a FLR <30% in normal livers, or 40% in livers chemotherapy damaged livers.
* 18 years and older
* Patients up to ECOG 3 (not more than 50% bedbound)
* Patients with non-resected primary colorectal cancer (CRC) may be included if and only if there is an intent to remove the CRC after the liver treatment (liver first approach)
* Staging CT chest and (if symptomatic) CT/MRI excludes unresectable extrahepatic disease, while metastatic disease that may be cured in the future, is included.
* Patients with resectable lung metastases or lung metastases that and be ablated can be included only after statement about resectability/ablatability by tumor board
* Patients have to be to understand the trial and provide informed consent.

Exclusion Criteria:

* Patients with extrahepatic disease other than lung metastases
* Patients with metastatic disease to the lung that cannot be ablated or resected will be excluded
* Patients with intrahepatic Cholangiocarcinoma (IHCC)
* Patients with Perihilar Cholangiocarcinoma (PHCC)
* Patients with Hepatocellular Carcinoma (HCC)
* Pregnant or lactating women will not be eligible
* Potential to get pregnant has to be excluded (obligatory contraception etc.)
* Progression by modified RECIST criteria on cross-sectional imaging after conversion chemotherapy is an exclusion criterion. Complete response in cross-sectional imaging after conversion chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Ability of each center to enroll 3 patients in 12 months without mortality due to the intervention. | 1 year/ 90 day mortality
  Ability of each center to enroll 3 patients for PVE/HVE in 12 months safely and perform the procedure including the liver resection without 90-day mortality after resection due to complications. If this goal is achieved center will be enrolled in DRAGON 2.

SECONDARY OUTCOMES:
Efficacy assessment: standardized future liver remnant volume | 6 weeks
  Increased of standardized future liver remnant volume between initial imaging and imaging at 1 week, 3 weeks, 6 weeks, degree of hypertrophy based on standard future liver remnant volume, kinetic growth
Feasibility assessment: resection rate | 1 year follow up
  ion of patients proceeding to complete resection (=resection rate)
Mortality assessment | 90 days
  90-mortality after resection
Overall survival after PVE/HVE | 1 year follow up
  Overall survival
Oncological effectiveness of PVE/HVE | 1 year
  Disease-free survival after 1 year
General complication assessment | 90 days
  90-day complications, general (Clavien-Dindo)
Liver specific complication assessment | 90 days
  90-day complications, liver specific (FABIB-classification)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M van Dam, MD PhD, Principal Investigator — Maastricht University Medical Center; Erik Schadde, MD FACS FEBS, Principal Investigator — Kantonsspital Winterthur/ Rush University Medical Center, Chicago; Marc AH Bemelmans, MD PhD, Principal Investigator — Maastricht University Medical Center; Christiaan van der Leij, MD PhD, Principal Investigator — Maastricht University Medical Center; Christoph A Binkert, Prof.Dr.Med, Principal Investigator — Cantonal Hospital Winterthur
Locations (42):
- United States (3):
  - Yale School of Medicine, New Haven, Connecticut
  - Rush University Medical Center, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Monash Health, Clayton, Clayton, Victoria
- Social Medical Center, South, Vienna, Austria
- Belgium (3):
  - Hôpital Erasme, Brussels, Brussels Capital
  - CHU-UCL Namur site Godinne, Yvoir, Namen
  - CHU de Liège, Liège
- Canada (2):
  - The Ottawa Hospital, Ottawa, Ontario
  - McGill University Health Center, Montreal
- Germany (3):
  - Klinikum Saarbrücken gGmbH, Saarbrücken, Saarland
  - University Hospital Halle (Saale), Halle, Saxony-Anhalt
  - Frankfurt University Hospital, Frankfurt
- Italy (4):
  - Policlinico Sant'Orsola-Malpighi, Bologna
  - Fondazione Poliambulanza, Brescia
  - IRCCS San Raffaele Hospital, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Netherlands (8):
  - Maastricht University Medical Center+, Maastricht, Limburg
  - Amsterdam UMC, location AMC, Amsterdam, North Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - Amsterdam Medical Centers, Location VUmc, Amsterdam
  - Amphia, Breda
  - Maxima Medisch Centrum, Eindhoven
  - University Medical Center Groningen, Groningen
  - Universitair Medisch Centrum Utrecht, Utrecht
- Oslo University Hospital, Oslo, Norway
- Spain (6):
  - University Hospital Germans Trias I Pujol, Badalona, Barcelona
  - University Hospital Parc Taulí, Sabadell, Barcelona
  - Hospital Universitari Mútua Terrassa, Terrassa, Barcelona
  - Hospital Universitari Dr. Josep Trueta, Girona, Gerona
  - Clínic de Barcelona, Barcelona
  - University Hospital Miguel Servet, Zaragoza
- Sweden (2):
  - Linköping University Hospital, Linköping
  - Karolinska University Hospital, Stockholm
- Switzerland (2):
  - Claraspital & Clarunis University Hospital Basel, Basel, Canton of Basel-City
  - Kantonsspital Winterthur (KSW), Winterthur
- United Kingdom (5):
  - University Hospital Southampton, Southampton, Hampshire
  - Aintree University Hospital, Liverpool, Merseyside
  - Belfast Health and Social Care Trust, Belfast
  - King's college hospital NHS foundation trust, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: Yes
upon reasonable request after publication.
Supporting Information: Study Protocol
Time Frame: Study protocol has already been published : https://pubmed.ncbi.nlm.nih.gov/35790566/
  Other information may be shared upon reasonable request after publication
URL: http://dragontrial.com

REFERENCES:
- [Derived] Korenblik R, James S, Smits J, Diaz-Nieto R, Davis R, Chan BKY, Erdmann JI, Zijlstra IAJ, Arntz PJW, Kollmar O, Hoffmann MH, Vass DG, Lindsay R, Serenari M, Cappelli A, Gobardhan PD, Imani F, Suarez YF, Munos FG, Grunhagen DJ, Moelker A, Pieterman KJ, Kleeff J, Wohlgemuth WA, Herrero E, Gelabert A, Breitenstein S, Seeger N, Detry O, Gerard L, Sandstrom PA, Bjornsson B, Aldrighetti LA, De Cobelli F, Leclercq WKG, van Baardewijk LJ, Croagh D, De Boo DW, Kingham TP, Ridouani F, Metrakos P, Valenti D, Kalil J, Fretland AA, Carling U, Martel G, Ryan S, Udupa V, Macdonald A, Tasse JC, Stavrou GA, Spuentrup E, Borobia FG, Criado E, Sparrelid E, Delle M, Navines-Lopez J, Moragues JS, Andorra EC, Schnitzbauer A, Vogl TJ, Heil J, Primrose JN, Modi S, Fouraschen SMG, Bokkers RPH, de Boer MT, Borel Rinkes IHM, Smits MLJ, Gruenberger T, Baclija I, Billingsley KG, Madoff DC, Serrablo A, Sarria L, Wang X, Xudong Q, Winkens B, Olde Damink SWL, Bemelmans MHA, Dewulf MJL, Binkert CA, Schadde E, van der Leij C, van Dam RM; DRAGON collaborative study group. Safety and efficacy of combined portal and hepatic vein embolisation in patients with colorectal liver metastases (DRAGON1): a multicentre, single-arm clinical trial. Lancet Reg Health Eur. 2025 Apr 10;53:101284. doi: 10.1016/j.lanepe.2025.101284. eCollection 2025 Jun. PMID 40255933
- [Derived] Korenblik R, Olij B, Aldrighetti LA, Hilal MA, Ahle M, Arslan B, van Baardewijk LJ, Baclija I, Bent C, Bertrand CL, Bjornsson B, de Boer MT, de Boer SW, Bokkers RPH, Rinkes IHMB, Breitenstein S, Bruijnen RCG, Bruners P, Buchler MW, Camacho JC, Cappelli A, Carling U, Chan BKY, Chang DH, Choi J, Font JC, Crawford M, Croagh D, Cugat E, Davis R, De Boo DW, De Cobelli F, De Wispelaere JF, van Delden OM, Delle M, Detry O, Diaz-Nieto R, Dili A, Erdmann JI, Fisher O, Fondevila C, Fretland A, Borobia FG, Gelabert A, Gerard L, Giuliante F, Gobardhan PD, Gomez F, Grunberger T, Grunhagen DJ, Guitart J, Hagendoorn J, Heil J, Heise D, Herrero E, Hess GF, Hoffmann MH, Iezzi R, Imani F, Nguyen J, Jovine E, Kalff JC, Kazemier G, Kingham TP, Kleeff J, Kollmar O, Leclercq WKG, Ben SL, Lucidi V, MacDonald A, Madoff DC, Manekeller S, Martel G, Mehrabi A, Mehrzad H, Meijerink MR, Menon K, Metrakos P, Meyer C, Moelker A, Modi S, Montanari N, Navines J, Neumann UP, Peddu P, Primrose JN, Qu X, Raptis D, Ratti F, Ridouani F, Rogan C, Ronellenfitsch U, Ryan S, Sallemi C, Moragues JS, Sandstrom P, Sarria L, Schnitzbauer A, Serenari M, Serrablo A, Smits MLJ, Sparrelid E, Spuntrup E, Stavrou GA, Sutcliffe RP, Tancredi I, Tasse JC, Udupa V, Valenti D, Fundora Y, Vogl TJ, Wang X, White SA, Wohlgemuth WA, Yu D, Zijlstra IAJ, Binkert CA, Bemelmans MHA, van der Leij C, Schadde E, van Dam RM. Dragon 1 Protocol Manuscript: Training, Accreditation, Implementation and Safety Evaluation of Portal and Hepatic Vein Embolization (PVE/HVE) to Accelerate Future Liver Remnant (FLR) Hypertrophy. Cardiovasc Intervent Radiol. 2022 Sep;45(9):1391-1398. doi: 10.1007/s00270-022-03176-1. Epub 2022 Jul 5. PMID 35790566